CLINICAL TRIAL: NCT02905149
Title: Impact of the Serratus Plane Block in Pain and the Use of Opioids in Breast
Brief Title: Impact of the Serratus Plane Block in Pain and the Use of Opioids in Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBMS-SPB
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2017-08

CONDITIONS: Surgery; Breast Reconstruction
Keywords: Oncological; Surgery; Breast; Reconstruction

STUDY DESIGN:
Intervention Model Description: Two group parallel arm. With study group receiving regional anesthestic block with levobupivacaine and control group receiving standard care with intravenous analgesia only
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serrato (Experimental): Standard anesthesia+serratus plane block.
  Interventions: Procedure: Serrato
- Control (Placebo Comparator): Standard anesthesia
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Serrato — Serratus plane block.
  Arms: Serrato
Procedure: Control — Standard anesthesia
  Arms: Control

SUMMARY:
The purpose of this project is to evaluate the analgesic efficacy of a regional anesthesia technique ( interfascial block at the serratus muscle) performed in patient undergoing breast surgery and the effect of this technique on postoperative analgesia.

DETAILED DESCRIPTION:
Regional analgesia techniques have shown to have benefits over conventional analgesia. The lower opioids analgesics requirements decrease side effects associated with the use of this type of medication. It is also increasingly established scientific evidence that reducing opioids administration may play a role in prognosis of cancer patients given the immunosuppressive effect of these drugs.

In patients undergoing oncologic/reconstructive breast surgery paravertebral block has been traditionally performed, however the paravertebral space lacks a clear anatomical barrier from the spinal cord so the drugs administered can diffuse to the intervertebral foramen causing deeper levels of blocks (epidural or spinal blocks) and injections at the paravertebral level are associated with serious complications both neurological and respiratory (meningitis, spinal hematomas abscesses, pneumothorax, respiratory failure. This has led to the development of less invasive technique with an improved safety profile.

The serratus plane block falls within the framework of these newly developed techniques and the present study aims to assess its role in the management of the patient undergoing cancer / reconstructive surgery.

Considering a decrease in postoperative morphine consumption of 40% and the average consumption of opioid after breast surgery under general anesthesia is 15 milligrams ( standard deviation 8 mg ) investigators calculated that with an alpha error 5% power 80 % 56 patients (28 per group) were required to achieve a significant result. In anticipation of possible loss of sample, 60 patients were recruited . Analysis will be performed by intention to treat.

Quantitative variables (opioid consumption, pain estimated by VAS scale) will be analyzed using mixed linear model adding a random variable for interindividual variability for pain threshold. If the data do not meet the criteria of normality the Mann-Whitney U test will be used. If the groups differ in preoperative variables. Investigators will make a multivariable analysis adjusting for these variables. The need for rescue analgesia over time is analyzed by Kaplan-Meier curve where the terminal state is the administration of the first dose of opioid postoperatively. The difference side effects (nausea, pruritus, apnea, urinary retention, ileus ) and complications IPO questionnaire and analyzed by chi-square test and Fisher exact test. Scheffe correction will be applied for multiple comparison. Missing data are excluded from analysis.

The study has planned data monitoring and auditing by the IIS la Fe according to AEMPS guidelines. Registries will be obtained from electronic medical records available for double check procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, undergoing oncological surgery and/or breast reconstruction surgery whose pathology and surgical intervention supose at least a 24 hours hospital admission

Exclusion Criteria:

* ASA Physical Status Classification System- IV.- Morbid obesity (Body mass index >40). -Impossibility of anatomical structures ultrasound identification in a satisfactory way (there can be no distinction in the interfascial plane between serratus and pectoral muscle). -Opioids treatment before surgery. Sepsis and/or infection at the puncture site.
* Haemostasis disorders. - Allergy to any of the drugs used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Mazzinari, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital de Manises, Manises, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazzinari G, Rovira L, Casasempere A, Ortega J, Cort L, Esparza-Minana JM, Belaouchi M. Interfascial block at the serratus muscle plane versus conventional analgesia in breast surgery: a randomized controlled trial. Reg Anesth Pain Med. 2019 Jan;44(1):52-58. doi: 10.1136/rapm-2018-000004. PMID 30640653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Serrato | Control
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serrato | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Usage
Description: Total opioid usage in the first 24 hours (intra and postoperative) (in morphine milligrmas, fentanyl/morphine conversion = 10 mcgs/1mg). Opioid used will be fentanyl and morphine. Fentanyl will be converted in morphine milligrams equivlents to caluclate the total first 24H dose.
Time Frame: First 24 hours after surgery
Population: 2 participants were lost to follow up because of malfunctioning of the electronic device administering the potoperative opioid
Measure: Median (95% Confidence Interval); unit: milligrams
Arm/Group | Serrato | Control
Number analyzed (Participants) | 28 | 30
milligrams | 18.5 [17 to 24] | 30 [26 to 35]
Statistical Analysis 1: Comparison: Serrato vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison; Median Difference (Final Values) = 9, 95% CI 2-sided [4 to 14.5] — Generalized Hodges-Lehmann median difference is used. These are robust to the possibility that the population distributions in the two groups are different in ways other than location. It may not represent the raw median difference

2. Secondary Outcome: Pain at Rest and Coughing
Description: Pain at rest and coughing at 24h postoperative (Visual analogue scale 0-10 with 0 meaning no pain and 10 meaning the worst imaginable pain). High score mean worse outcomes
Time Frame: First 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Serrato | Control
Number analyzed (Participants) | 28 | 30
units on a scale
  Worst pain in 24h | 4 [3 to 6] | 6 [4 to 8]
  Least pain in 24h | 0 [0 to 0] | 0 [0 to 2]
  Pain interf. with activities in bed | 1 [0 to 3] | 1 [0 to 6]
  Pain interf. with breathing or coughing | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Time to First Opioid Administration on the Ward
Description: Time to first opioid administration on the ward
Time Frame: First 24 hours after surgery
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Serrato | Control
Number analyzed (Participants) | 28 | 30
hours | 7.95 [4.61 to 11.28] | 2.9 [0.8 to 5]

4. Secondary Outcome: Presence of Opioid Related Complications
Description: presence of nausea/vomit or apnea or urinary retention or ileus is assessed. It is a dicothomic composite (yes or no).
Time Frame: First 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Serrato | Control
Number analyzed (Participants) | 28 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours after surgery
Arm/Group | Serrato | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The blinding method cannot entirely exclude ascertainment bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT02905149/Prot_SAP_000.pdf